CLINICAL TRIAL: NCT06840405
Title: Cortical Activation During Forward and Backward Walking in Individuals With Chronic Stroke
Brief Title: Cortical Activation During Walking in Stroke
Status: Recruiting | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU113210AF1
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Forward walking; Backward walking; Brain activity; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After stroke, damage to one cerebral hemisphere disrupts the normal balance of activity between the two hemispheres. The affected hemisphere typically exhibits reduced excitability, whereas the unaffected side may demonstrate increased excitability. This phenomenon, referred to as interhemispheric imbalance, further inhibits activity in the affected hemisphere, thereby restricting motor recovery. According to the interhemispheric competition model, enhancing excitability in the affected hemisphere and/or suppressing excitability in the unaffected hemisphere may contribute to the improvement of motor function in individuals with stroke. Furthermore, as motor function recovers, the balance of interhemispheric activation in motor-related cortical areas undergoes corresponding changes. Previous studies have shown that treadmill training enhances the excitability of the primary motor cortex in both hemispheres of stroke patients, as well as increases excitability across multiple cortical and subcortical regions in both hemispheres. However, it remains unclear whether treadmill training can normalize the interhemispheric imbalance in stroke patients. Additionally, the effects of forward and backward walking on the activity of motor-related brain regions in individuals with stroke are still unclear. Therefore, this cross-sectional study aims to investigate the changes in motor-related brain activity during forward walking and backward walking in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months after the diagnosis of stroke
* Independent walking over at least 7m with or without a walking aid
* Mini-mental state examination score ≥ 24

Exclusion Criteria:

* Had difficulty in backward walking
* Any neuromuscular disorders history
* With visual or auditory disorders
* Unstable cardiac status or uncontrolled hypertension
* Any musculoskeletal disorders that would affect walking ability

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic stroke
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Brain activity | One-time measurement during a one-minute walking task at a single study visit
  Using functional near infrared spectroscopy to measure the oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) in the bilateral prefrontal cortex, supplementary motor area and primary motor cortex.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No